CLINICAL TRIAL: NCT04907851
Title: A Modular, Phase II, Open-Label, Multicentre Study to Assess the Preliminary Efficacy and Safety of RXC004, in Patients With Advanced Solid Tumours That Have Progressed Following Therapy With Current Standard of Care
Brief Title: A Study to Assess RXC004 Efficacy in Advanced Solid Tumours After Progression on Standard of Care (SoC) Therapy (PORCUPINE2)
Acronym: KEYNOTE-E86
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Redx Pharma Ltd (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RXC004/0003; MK-3475-E86 (Other: Collaboration requirements); KEYNOTE-E86 (Other: Collaboration requirements); 2020-005804-20 (EudraCT Number)
Record Dates: First submitted 2021-05-25; First posted 2021-06-01 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumours
Keywords: Open-Label; RXC004; Ring finger protein 43; Pancreatic ductal adenocarcinoma; Biliary tract cancer; Efficacy; Safety; Pharmacokinetics; Pancreatic cancer; Cholangiocarcinoma; Gallbladder; Ampullary Cancer; Ampulla of Vater; MK-3475-E86; zamaporvint
MeSH Terms: conditions — Biliary Tract Neoplasms; Pancreatic Neoplasms; Cholangiocarcinoma | interventions — Denosumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Module 1 - RNF43 Mutated Advanced (unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) (Experimental): Patients (Karnofsky performance status ≥70) will be recruited and dosed with RXC004 (2 mg once daily [QD], orally) within 6 weeks of progression following 1st line SoC treatment.
  Interventions: Drug: RXC004; Biological: Denosumab
- Module 2 -Advanced (unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) (Experimental): Patients (Eastern Cooperative Oncology Group [ECOG] performance status 0-1) will be recruited and dosed with RXC004 within 6 weeks of progression, following 1st line SoC treatment.
  Interventions: Drug: RXC004; Biological: Denosumab
- Module 3-Advanced (unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy (Experimental): Patients (ECOG performance status 0-1) will be recruited and dosed with RXC004 (1.5 mg QD, orally) in combination with pembrolizumab 400 mg IV infusion every 6 weeks (q6w) within 6 weeks of progression, following 1st line Soc treatment.
  Interventions: Drug: RXC004; Biological: Denosumab; Biological: pembrolizumab

INTERVENTIONS:
Drug: RXC004 — RXC004 will be administered orally, 2 mg QD; Dose Formulation: 0.5 mg or 1 mg capsules.
  Other Names: zamaporvint
  Arms: Module 1 - RNF43 Mutated Advanced (unresectable)/Metastatic Pancreatic Cancer (Stage III/IV)
Drug: RXC004 — RXC004 will be administered orally, 2 mg QD (Cohort 1, Module 2) and 1 mg QD (Cohort 2, Module 2); Dose Formulation: 0.5 mg or 1 mg capsules.
  Other Names: zamaporvint
  Arms: Module 2 -Advanced (unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV)
Drug: RXC004 — RXC004 will be administered orally, 1.5 mg QD; Dose Formulation: 0.5 mg or 1 mg capsules.
  Other Names: zamaporvint
  Arms: Module 3-Advanced (unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Biological: Denosumab — Denosumab will be administered via subcutaneous (SC) injection, 120 mg once every month; Use: Prophylactic
Biological: pembrolizumab — Pembrolizumab will be administered via intravenous infusion, 400 mg dose once every 6 weeks
  Other Names: KEYTRUDA®
  Arms: Module 3-Advanced (unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy

SUMMARY:
This study is to evaluate the preliminary efficacy and safety of RXC004 monotherapy and in combination with pembrolizumab in advanced solid tumours that have progressed following SoC treatment.

DETAILED DESCRIPTION:
This Phase II, modular, open label, multicentre study initially opened with ring finger protein 43 (RNF43) loss of function (LoF) mutation-positive pancreatic ductal adenocarcinoma (PDAC) (Module 1) and molecularly unselected biliary tract cancer (BTC) (Module 2) modules. Module 3 will investigate RXC004 in combination with pembrolizumab in BTC. Modules 1 and 2 are monotherapies and Module 3 is the combination therapy.

The primary objective of the study is to assess the preliminary efficacy of RXC004 in each module. This will be evaluated in terms of progression free survival (PFS) at 6 months in Modules 1 and 2, and in terms of Objective response rate (ORR) in Module 3. Following radiological progression, patients will be followed-up for survival.

ELIGIBILITY:
Core Inclusion Criteria:

* At least one lesion that is measurable by RECIST 1.1 at baseline (within 6 weeks prior to start of study treatment).
* Mandatory paired biopsies; Patients must have at least one lesion suitable for biopsy at screening
* Adequate organ and marrow function
* Female patients of childbearing potential must have a negative pregnancy test prior to start of dosing
* Female patients of childbearing potential and male patients with female partners of childbearing potential must agree to use a highly effective method of contraception during the study from the time of treatment initiation, and for at least 5 months after the last dose of study drug.

Module 1 (PDAC) Specific Inclusion Criteria

* Histological documentation of advanced (unresectable)/metastatic (Stage III/IV) PDAC, with documented loss of function tumour mutation in RNF43
* Patients must have received one prior systemic treatment for advanced (unresectable)/metastatic PDAC (Stage III/IV), with clear evidence of radiological disease progression
* Patients must be enrolled and receive first dose of study treatment within 6 weeks of radiologically confirmed progression
* Karnofsky performance status ≥70.

Module 2 and Module 3 (BTC) Specific Inclusion Criteria

* Histological documentation of advanced (unresectable)/metastatic (Stage III/IV) BTC (intrahepatic or extrahepatic cholangiocarcinoma, ampulla of Vater, or gallbladder cancer)
* Patients must have received one prior systemic treatment for advanced (unresectable)/metastatic BTC, with clear evidence of radiological disease progression
* Patients must be enrolled and receive first dose of study treatment within 6 weeks of radiologically confirmed progression
* ECOG status 0 or 1.

Core Exclusion Criteria:

* Prior therapy with a compound of the same mechanism of action as RXC004
* Patients at higher risk of bone fractures
* Any known uncontrolled inter-current illness or persistent clinically significant toxicity related to prior anti-cancer treatment
* Patients who have any history of an active (requiring treatment) other malignancy within 2 years of study entry
* Patients with known or suspected brain metastases
* Use of anti-neoplastic agents
* Patients with a known hypersensitivity to any RXC004 excipients
* Patients with a contra-indication for denosumab treatment
* Patients who are pregnant or breast-feeding
* Known active human immunodeficiency viruses (HIV), hepatitis B (HBV), or hepatitis C (HCV) infections
* Use of any live or live-attenuated vaccines against infectious diseases (e.g., influenza nasal spray, varicella) within 4 weeks (28 days) of initiation of study treatment
* Mean resting corrected QTcF >470 ms, obtained from triplicate ECGs performed at screening.

There are no exclusion criteria specific to Modules 1 and 2.

Module 3 Specific Exclusion Criteria:

* Patients with any contraindication to the use of pembrolizumab as per approved label
* Has received prior therapy with an anti-programmed cell death-1 (anti-PD-1), anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor, and was discontinued from that treatment due to a Grade 3 or higher AE
* Has received prior radiotherapy within 2 weeks of start of study treatment or have had a history of radiation pneumonitis
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of pembrolizumab in this study
* Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease
* Has an active infection requiring systemic therapy
* Patients with a history of allogeneic tissue/solid organ transplant
* Patients with active infections, including tuberculosis, HIV, HBV, or HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Australia (2):
  - Wollongong Hospital, Wollongong, New South Wales
  - The Alfred Hospital - Alfred Health, Melbourne, Victoria
- United Kingdom (11):
  - Cambridge University Hospital NHS Foundation Trust, Cambridge
  - Beatson West of Scotland Cancer Care, Glasgow
  - St James University Hospital, Leeds
  - Barts Cancer Institute - Haemato-Oncology, London
  - University College Hospitals NHS Foundation Trust, London
  - Royal Free London Foundation NHS Trust, London
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital, London
  - The Christie NHS Foundation Trust - Medical Oncology, Manchester
  - Oxford Cancer and Haematology Centre Churchill Hospital, Oxford
  - Weston Park Hospital, Sheffield
  - The Royal Marsden Hospital (Surrey), Sutton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 10 December 2021 to 22 Nov 2023 at multiple centers in Australia, and United Kingdom.
Pre-assignment Details: Patients who met the inclusion criteria, and none of the exclusion criteria were enrolled to the study. All study assessments were performed as per the Schedule of Assessment.
Groups:
- Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV): Patients (Karnofsky performance status ≥70) were recruited and dosed with RXC004 (2 mg once daily [QD] orally) within 6 weeks of progression following 1st line Standard of Care (SoC) treatment.
- Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV): Patients (Eastern Cooperative Oncology Group [ECOG] performance status 0-1) were recruited and dosed with RXC004 within 6 weeks of progression following 1st line SoC treatment.
- Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy: Patients (ECOG performance status 0-1) were recruited and dosed with RXC004 (1.5 mg QD orally) in combination with pembrolizumab 400 mg IV infusion every 6 weeks (q6w) within 6 weeks of progression following 1st line SoC treatment.
Period: Overall Study
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Started | 6 | 20 | 19
Completed | 0 | 3 | 9
Not Completed | 6 | 17 | 10
Not completed — Consent withdrawn | 1 | 2 | 0
Not completed — Death | 5 | 15 | 10

BASELINE CHARACTERISTICS:
Population: Full analysis set included all patients who were enrolled and received at least one dose of RXC004 in Modules 1 and 2, and at least one dose of RXC004 or pembrolizumab in Module 3.
Groups:
- Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV): Patients (Karnofsky performance status ≥70) were recruited and dosed with RXC004 (2 mg QD orally) within 6 weeks of progression following 1st line SoC treatment.
- Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV): Patients (ECOG performance status 0-1) were recruited and dosed with RXC004 within 6 weeks of progression following 1st line SoC treatment.
- Total: Total of all reporting groups
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy | Total
Number analyzed (Participants) | 6 | 20 | 19 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (7.94) | 55.8 (14.72) | 58.1 (10.85) | 58.1 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 12 | 25
  Male | 3 | 10 | 7 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 0 | 2
  Black or African American | 0 | 0 | 2 | 2
  White | 3 | 19 | 17 | 39
  Other | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 5 | 17 | 19 | 41
  Not Stated | 0 | 1 | 0 | 1
  Unknown | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Monotherapy (Modules 1 and 2): Progression Free Survival Rate at 6 Months
Description: The anti-tumour activity of RXC004 was assessed. Progression free survival rate at 6 months was defined as the percentage of patients who remained alive and free of progression at 6 months according to Kaplan-Meier estimates.
Time Frame: At 6 months
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV)
Number analyzed (Participants) | 6 | 20
percentage of participants | NA [NA to NA] — The estimate of PFS at 6-months could not be calculated as the final surviving patient withdrew consent and was censored at 2.73 months. The Kaplan-Meier survival curve, from which the estimates would have been derived, did not extend to 6-months. | 6.1 [0.73 to 20.53]

2. Primary Outcome: Combination Therapy (Module 3): Objective Response Rate (ORR)
Description: The anti-tumour activity of RXC004 as a combination therapy was assessed. ORR was defined as the percentage of patients with a best overall response of complete response or partial response based on local investigator assessment as defined in RECIST 1.1.
Time Frame: Up to 23 months
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy: Patients (ECOG performance status 0-1) were recruited and dosed with RXC004 (1.5 mg QD orally) in combination with pembrolizumab 400 mg IV infusion q6w within 6 weeks of progression following 1st line SoC treatment.
Arm/Group | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Number analyzed (Participants) | 19
percentage of participants | 0 [0.00 to 14.59]

3. Secondary Outcome: Monotherapy (Modules 1 and 2): ORR
Description: The preliminary efficacy of RXC004 was assessed. ORR was defined as the percentage of patients with a best overall response of complete response (CR) or partial response (PR) based on local Investigator assessment as defined in RECIST 1.1.
Time Frame: Up to 23 months
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV)
Number analyzed (Participants) | 6 | 20
percentage of participants | 16.7 [0.85 to 58.18] | 5.0 [0.26 to 21.61]

4. Secondary Outcome: Monotherapy (Modules 1 and 2) and Combination Therapy (Module 3): Disease Control Rate (DCR)
Description: The preliminary efficacy of RXC004 as a monotherapy and as a combination therapy was assessed. DCR was defined as the percentage of patients with a best overall response of either CR, PR or stable disease (SD) for at least 6 weeks.
Time Frame: Up to 23 months
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV): Patients (Karnofsky performance status≥70) were recruited and dosed with RXC004 (2 mg QD orally) within 6 weeks of progression following 1st line SoC treatment.
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Number analyzed (Participants) | 6 | 20 | 19
percentage of participants | 16.7 [0.85 to 58.18] | 25.0 [10.41 to 45.56] | 31.6 [14.75 to 53.00]

5. Secondary Outcome: Monotherapy (Modules 1 and 2) and Combination Therapy (Module 3): PFS
Description: The preliminary efficacy of RXC004 as a monotherapy and as a combination therapy was assessed. PFS was defined as the time from first dose of study treatment until the date of disease progression or death (by any cause in the absence of progression) regardless whether the patient withdrew from the assigned study treatment or received another anticancer prior to progression.
Time Frame: Up to 23 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV): Patients (ECOG performance status 0-1) were recruited and dosed with RXC004 within 6 weeks of progression following1st line SoC treatment.
- Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy: Patients (ECOG performance status 0-1) were recruited and dosed with RXC004(1.5 mg QD orally) in combination with pembrolizumab 400 mg IV infusion q6w within 6 weeks of progression following 1st line SoC treatment.
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Number analyzed (Participants) | 6 | 20 | 19
months | 1.4 [0.72 to NA] — Due to insufficient number of participants with events, estimates were not calculable using methodology specified in SAP. | 1.4 [1.38 to 2.04] | 1.41 [1.41 to 2.53]

6. Secondary Outcome: Monotherapy (Modules 1 and 2) and Combination Therapy (Module 3): Best Percentage Change in Tumor Size
Description: The preliminary efficacy of RXC004 as a monotherapy and as a combination therapy was assessed. The best percentage change in tumour size was determined at a patient level. For each patient, it represents the largest decrease (or smallest increase) in tumour size. Percentage change in tumour size was derived at each visit by the percentage change from baseline in the sum of diameters of all target lesions.
Time Frame: Up to 23 months
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Percentage change in tumour size
Groups:
- Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy: Patients (ECOG performance status 0-1) were recruited and dosed with RXC004(1.5 mg QD orally) in combination with pembrolizumab 400 mg IV infusion q6wwithin 6 weeks of progression following 1st line SoC treatment.
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Number analyzed (Participants) | 5 | 20 | 17
Percentage change in tumour size | 41.67 [-57.1 to 93.2] | 20.06 [-78.8 to 87.9] | 30.61 [-33.3 to 61.3]

7. Secondary Outcome: Monotherapy (Modules 1 and 2) and Combination Therapy (Module 3): Overall Survival (OS)
Description: The preliminary efficacy of RXC004 as a monotherapy and as a combination therapy was assessed. OS was defined as the time from first day of study treatment until death due to any cause.
Time Frame: Up to 23 months
Population: Full Analysis Set included all patients who enrolled and received at least one dose of RXC004 in Modules 1 and 2, and at least one dose of RXC004 or pembrolizumab in Module 3.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Number analyzed (Participants) | 6 | 20 | 19
Months | 5.3 [0.7 to NA] — Due to insufficient number of participants with events, estimates were not calculable using methodology specified in SAP. | 7.1 [3.5 to 13.6] | 4.7 [2.9 to NA] — Due to insufficient number of participants with events, therefore data was not calculated as per methodology specified in SAP.

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: The pharmacokinetics (PK) of RXC004 as a monotherapy and as a combination therapy was assessed.
Time Frame: At Cycle 0 Day 1 and Cycle 1 Day 15 (Each cycle was 21 days in length)
Population: PK Analysis Set included all patients in the safety analysis set who have had at least one blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Number analyzed (Participants) | 6 | 17 | 16
nanogram per milliliter (ng/mL)
  Cycle 0 Day 1: number analyzed (Participants) | 6 | 16 | 15
  Cycle 0 Day 1 | 107 (31.4) | 78.7 (43.9) | 57.6 (44.1)
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 17 | 16
  Cycle 1 Day 15 | 140 (50.8) | 99.5 (50.7) | 67.5 (56.8)

9. Secondary Outcome: Time to Cmax (Tmax)
Description: The PK (tmax) of RXC004 as a monotherapy and as a combination therapy was assessed.
Time Frame: At Cycle 0 Day 1 and Cycle 1 Day 15 (Each cycle was 21 days in length)
Population: PK Analysis Set included all patients in the safety analysis set who have had at least one blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Number analyzed (Participants) | 6 | 17 | 16
hour (h)
  Cycle 0 Day 1: number analyzed (Participants) | 6 | 16 | 15
  Cycle 0 Day 1 | 1.49 (36.3) | 1.44 (51.3) | 1.66 (45.9)
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 17 | 16
  Cycle 1 Day 15 | 1.49 (36.3) | 1.44 (51.3) | 1.66 (45.9)

10. Secondary Outcome: Minimum Observed Concentration Across the Dosing Interval (Cmin)
Description: The PK (Cmin) of RXC004 as a monotherapy and as a combination therapy was assessed.
Time Frame: At Cycle 1 Day 15 (The cycle was 21 days in length) (Up to 23 months)
Population: PK Analysis Set included all patients in the safety analysis set who have had at least one blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Number analyzed (Participants) | 5 | 17 | 16
ng/mL | 22.0 (37.5) | 19.5 (110) | 9.79 (153)

11. Secondary Outcome: Terminal Rate Constant (λz)
Description: The PK (λz) of RXC004 as a monotherapy and as a combination therapy was assessed.
Time Frame: At Cycle 0 Day 1 (The cycle was 21 days in length)
Population: PK Analysis Set included all patients in the safety analysis set who have had at least one blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: one per hour (1/h)
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Number analyzed (Participants) | 6 | 16 | 15
one per hour (1/h) | 0.0660 (36.5) | 0.0660 (32.4) | 0.0655 (28.0)

12. Secondary Outcome: Terminal Half-life (t½)
Description: The PK (t½) of RXC004 as a monotherapy and as a combination therapy was assessed.
Time Frame: At Cycle 0 Day 1(The cycle was 21 days in length)
Population: PK Analysis Set included all patients in the safety analysis set who have had at least one blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Number analyzed (Participants) | 6 | 16 | 15
hour (h) | 10.5 (36.5) | 9.90 (27.6) | 10.6 (29.0)

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to Infinity (AUC0-∞)
Description: The PK (AUC0-∞) of RXC004 as a monotherapy and as a combination therapy was assessed.
Time Frame: At Cycle 0 Day 1 (The cycle was 21 days in length)
Population: PK Analysis Set included all patients in the safety analysis set who have had at least one blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Number analyzed (Participants) | 6 | 16 | 15
hour*nanogram per milliliter (h*ng/mL) | 891 (21.8) | 690 (43.5) | 511 (47.0)

14. Secondary Outcome: Total Plasma Clearance After Oral Administration (CL/F)
Description: The PK(CL/F) of RXC004 as a monotherapy and as a combination therapy was assessed.
Time Frame: At Cycle 0 Day 1 (The cycle was 21 days in length)
Population: PK Analysis Set included all patients in the safety analysis set who have had at least one blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per hour (mL/h)
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Number analyzed (Participants) | 6 | 16 | 15
milliliter per hour (mL/h) | 2250 (21.8) | 2900 (43.5) | 2940 (47.0)

15. Secondary Outcome: Apparent Volume of Distribution After Oral Administration (Vz/F)
Description: The PK (Vz/F) of RXC004 as a monotherapy and as a combination therapy was assessed.
Time Frame: At Cycle 0 Day 1 (The cycle was 21 days in length)
Population: PK Analysis Set included all patients in the safety analysis set who have had at least one blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter (mL)
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Number analyzed (Participants) | 6 | 16 | 15
milliliter (mL) | 29700 (28.9) | 41400 (31.0) | 44800 (40.4)

16. Secondary Outcome: Number of Patients With Adverse Events (AEs)
Description: The safety, and tolerability profile of RXC004 as a monotherapy and as a combination therapy was assessed. The grading scales found in the revised National Cancer Institute CTCAE latest version was utilized for all events with an assigned CTCAE grading. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL; Grade 4: Life-threatening, urgent intervention required; Grade 5: Death related to AE.
Time Frame: From time of signature of main study informed consent form throughout the treatment period and until the 30 days after last dose of RXC004 (Up to 23 months)
Population: Safety Set included all patients who enrolled and received at least one dose of RXC004 in Modules 1 and 2, and at least one dose of RXC004 or pembrolizumab in Module 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
Number analyzed (Participants) | 6 | 20 | 19
Participants
  Treatment-Emergent Adverse Event (TEAE) | 6 | 20 | 19
  Related TEAE | 4 | 17 | 18
  Grade >=3 TEAE | 4 | 8 | 10
  Related grade>=3 TEAE | 1 | 3 | 5
  Serious TEAE | 3 | 6 | 11
  Related Serious TEAE | 0 | 1 | 4
  TEAE leading to death | 0 | 0 | 1
  TEAE leading to permanent discontinuation or reduction or interruption of RXC004 | 3 | 10 | 11
  TEAE leading to permanent discontinuation of RXC004 | 1 | 2 | 6
  TEAE leading to reduction of RXC004 | 0 | 2 | 1
  TEAE leading to interruption of RXC004 | 0 | 9 | 7
  TEAE leading to permanent discontinuation or 0 6 interruption of Pembrolizumab | 0 | 0 | 6
  TEAE leading to permanent discontinuation of 0 5 Pembrolizumab | 0 | 0 | 5
  TEAE leading to interruption of Pembrolizumab | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From time of signature of main study informed consent form throughout the treatment period and until the 30 days after last dose of RXC004 (Up to 23 months)].
Description: Safety Set included all patients who enrolled and received at least one dose of RXC004 in Modules 1 and 2, and at least one dose of RXC004 or pembrolizumab in Module 3.
  All the AEs from Screening till study termination have been presented here before, and after receiving treatment.
Arm/Group | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy
All-Cause Mortality (participants affected / at risk) | 5/6 | 15/20 | 10/19
Serious Adverse Events (participants affected / at risk) | 3/6 | 6/20 | 11/19
Other Adverse Events (participants affected / at risk) | 6/6 | 20/20 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) (N=6) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) (N=20) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy (N=19)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (3)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Stoma site abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lacunar stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Module 1-RNF43 Mutated Advanced (Unresectable)/Metastatic Pancreatic Cancer (Stage III/IV) (N=6) | Module 2-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage III/IV) (N=20) | Module 3-Advanced (Unresectable)/Metastatic Biliary Tract Cancer (Stage Ill/IV) Combination Therapy (N=19)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (8) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 8 (9) | 6 (8)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 10 (11) | 5 (5)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 3 (3)
Weight decreased (Investigations) | 1 (1) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 6 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 4 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 5 (5) | 13 (14) | 12 (13)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (6)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 13 (14) | 5 (5)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Steatorrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 9 (9) | 8 (9)
Pyrexia (General disorders) | 0 (0) | 4 (4) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 2 (2)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasal herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (3) | 4 (6)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arachnoid cyst (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT04907851/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT04907851/SAP_001.pdf